CLINICAL TRIAL: NCT06575114
Title: COVID-19 Vaccination Willingness in Older Adults Based on Self-determination Theory
Acronym: CVWIOABOSDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jing-Shan Deng (Other)
Responsible Party: Sponsor-Investigator, Jing-Shan Deng, Main responsibility and supervision, Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Organization: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K20230832
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Old Age; Debility; Vaccine Hesitancy; Vaccine Refusal
Keywords: Basic psychological needs; booster dose; COVID-19 vaccine; older adults; SARS-CoV-2; self-determination theory; willingness
MeSH Terms: conditions — Frailty; Vaccination Hesitancy; Vaccination Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: traditional health education (Other): In the control group, a conventional intervention will be used, and health education brochures on the COVID-19 vaccine will be distributed for the study participants to read on their own time. The contents of the brochure included basic knowledge concerning the SARS-CoV-2 coronavirus, COVID-19 vaccine, herd immunity, and precautions for vaccination.
  Interventions: Other: Self-determination theory-based health education measures
- Intervention group: Self-determination theory-based health education measures (Other): The intervention group will receive self-determination theory-based interventions, with targete interventions proposed based on the self-determination theory-including health-related talks and sharing sessions. To ensure that older individuals with varying levels of literacy understood the intervention, the process will be conducted in the local native dialect.
  Interventions: Other: Self-determination theory-based health education measures

INTERVENTIONS:
Other: Self-determination theory-based health education measures — In the control group, a conventional intervention will be used, and health education brochures on the COVID-19 vaccine will be distributed for the study participants to read on their own time. The intervention group will receive self-determination theory-based interventions, with targete interventions proposed based on the self-determination theory-including health-related talks and sharing sessions. To ensure that older individuals with varying levels of literacy understood the intervention, the process will be conducted in the local native dialect.
  Other Names: traditional health education

SUMMARY:
Introduction: The COVID-19 vaccine is an effective measure for preventing and controlling COVID-19 epidemics, and the World Health Organization lists older adults as a high-priority group for COVID-19 vaccination. However, the willingness of older people to be vaccinated against COVID-19 remains an important issue in achieving herd immunity. We investigated the effectiveness of a COVID-19 vaccine intervention for older adults, based on self-determination theory.

Methods and analysis: Questionnaires were administered to assess vaccine willingness at baseline and at 6 weeks following educational intervention programs concerning vaccination against COVID-19. Four nursing homes with a population size of over 100 will be selected and randomized into intervention and control groups. The control group will undergo conventional intervention methods, and the intervention group will undergo a comprehensive intervention program based on self-determination theory.

Ethics and dissemination: The study has been approved by the Ethics Committee of Taizhou Hospital, Zhejiang Province, China (approval number: K20230832).

DETAILED DESCRIPTION:
1. Study design and data collection This class pilot study will be conducted in September 2023 at a nursing home in Taizhou, China. This study has been approved by the Ethics Committee of Taizhou Hospital, Zhejiang Province, China (approval number: K20230832). All procedures will be performed in accordance with the guidelines of our institutional ethics committee and in compliance with the Declaration of Helsinki. The respondents' information will remain anonymous.
2. Patients and public involvement The study participants will be not involved in the design, implementation, or reporting of the study.

2.1 Recruitment 2.2.1 Inclusion criteria

1. 60 years old or above
2. Have not been vaccinated for COVID-19 or have not completed the fourth booster shot of the COVID-19 vaccine
3. Able to communication and willing to participate in the survey voluntarily 2.2.2 Exclusion criteria

(1) People with contraindications to vaccination (2) People with communication disorders (3) Those who do not want to participate in the survey 2.3.3 Grouping of study participants We will select four senior care institutions in Taizhou City with a population of 100 or more residents. We will divide them into intervention and control groups.

2.4 Sample size The sample size was determined using G*Power software v3.1.9.2 (Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany). It will be estimated for repeated measures between the two groups at a significance level of 0.05, effect size of 0.19, and power of 95%. The final calculated sample size is 182 participants. Assuming a 10% attrition rate over the course of the intervention, we set a target of recruiting 200 participants. Based on the number of repeated measurements, this represented 100 participants in each group.

2.5 Composition of investigators

1. One master's degree in public health
2. Four master's degrees in infection
3. Two physicians in infectious diseases
4. Two trained locals 2.6 Intervention 2.6.1 Control group: traditional health education In the control group, a conventional intervention will be used, and health education brochures on the COVID-19 vaccine will be distributed for the study participants to read on their own time. The contents of the brochure included basic knowledge concerning the SARS-CoV-2 coronavirus, COVID-19 vaccine, herd immunity, and precautions for vaccination.

2.6.2 Self-determination theory-based health education measures The intervention group received self-determination theory-based interventions, with targeted interventions proposed based on the self-determination theory-including health-related talks and sharing sessions. To ensure that older individuals with varying levels of literacy understood the intervention, the process was conducted in the local native dialect. Health lectures will be conducted to elicit and acknowledge the perspectives and emotions of our cohort of older adults toward vaccination, support their choices and initiatives, and provide a rationale for vaccination-related recommendations while communicating with them to better understand their major barriers toward vaccination. This will be done with the idea of meeting the autonomy and competence needs of our cohort, based on one of the basic premises of self-determination theory. Health-related lectures empower older adults to make autonomous decisions through cognitive reframing . It has been found that successful vaccination planning relies on people acquiring appropriate and adequate health-related knowledge. The three basic psychological needs of older adults will be met through communication and interaction, both with them and with significant members of their lives (e.g., caregivers, family members, doctors, and nurses) during sharing communication sessions. We also will seek to motivate the participants by asking them questions and awarding them gifts during each health lecture and sharing session. Competence needs will be met by developing challenges for our participant cohort . The entire intervention will last 6 weeks, and will be followed by a face-to-face questionnaire.

ELIGIBILITY:
Inclusion Criteria:

(1) ≥ 60 years of age; (2) had not previously been vaccinated with a COVID-19 vaccine, or had not yet received their fourth booster dose of the vaccine; and (3) had the ability to communicate verbally and volunteered to participate in the survey.

Exclusion Criteria:

(1) contraindications to vaccination; (2) communication disorders; and (3) unwillingness to participate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Willingness to vaccinate | 6 weeks
  Changes in Vaccination Wiilingness Scores for the Elderly

SECONDARY OUTCOMES:
Basic psychological needs | 6 weeks
  Changes in Basic psychological needs Scores for the Elderly
Vaccine literacy | 6 weeks
  Changes in Vaccine literacy Scores for the Elderly

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Shan Deng, postgraduate, Principal Investigator — Jing-Shan Deng WenZhou Medical University
Locations (1):
- Taizhou Hospital, Taizhou, Linhai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patrick H, Williams GC. Self-determination theory: its application to health behavior and complementarity with motivational interviewing. Int J Behav Nutr Phys Act. 2012 Mar 2;9:18. doi: 10.1186/1479-5868-9-18. PMID 22385676
- [Result] Silva MN, Markland D, Minderico CS, Vieira PN, Castro MM, Coutinho SR, Santos TC, Matos MG, Sardinha LB, Teixeira PJ. A randomized controlled trial to evaluate self-determination theory for exercise adherence and weight control: rationale and intervention description. BMC Public Health. 2008 Jul 9;8:234. doi: 10.1186/1471-2458-8-234. PMID 18613959
- [Result] Dube E, Gagnon D, Ouakki M, Bettinger JA, Guay M, Halperin S, Wilson K, Graham J, Witteman HO, MacDonald S, Fisher W, Monnais L, Tran D, Gagneur A, Guichon J, Saini V, Heffernan JM, Meyer S, Driedger SM, Greenberg J, MacDougall H; Canadian Immunization Research Network. Understanding Vaccine Hesitancy in Canada: Results of a Consultation Study by the Canadian Immunization Research Network. PLoS One. 2016 Jun 3;11(6):e0156118. doi: 10.1371/journal.pone.0156118. eCollection 2016. PMID 27257809
- [Result] Ntoumanis N, Ng JYY, Prestwich A, Quested E, Hancox JE, Thogersen-Ntoumani C, Deci EL, Ryan RM, Lonsdale C, Williams GC. A meta-analysis of self-determination theory-informed intervention studies in the health domain: effects on motivation, health behavior, physical, and psychological health. Health Psychol Rev. 2021 Jun;15(2):214-244. doi: 10.1080/17437199.2020.1718529. Epub 2020 Feb 3. PMID 31983293
- [Result] Gillison FB, Rouse P, Standage M, Sebire SJ, Ryan RM. A meta-analysis of techniques to promote motivation for health behaviour change from a self-determination theory perspective. Health Psychol Rev. 2019 Mar;13(1):110-130. doi: 10.1080/17437199.2018.1534071. Epub 2018 Oct 16. PMID 30295176